CLINICAL TRIAL: NCT00448045
Title: Prevention of Long-Term Respiratory Complications of Spinal Cord Injury: a Randomized Controlled Trial
Brief Title: Preventing Pneumonia and Other Respiratory Problems in Persons With Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Trevor Dyson-Hudson, M.D., Interim-Director, Spinal Cord Injury Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H133N060022
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injuries; Cough; Peak cough flow; Respiratory therapy; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Cough

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual and mechanical assisted cough (Experimental): Individuals will be given a pulse oximeter and taught both manually assisted and mechanically assisted coughing techniques to maximize their cough peak flow. Manually assisted coughing consists of air stacking to deep insufflations. An abdominal thrust is then applied upon glottic opening to augment the cough peak flow. Subjects will also have rapid access to a mechanical in-exsufflator (CoughAssistTM) and will be trained on how to access and use this device. Mechanically assisted coughing (MAC) involves the use of the CoughAssistTM to expand the lungs and then quickly reverse the pressure to rapidly empty the lungs with expiratory (cough) flows of 600 L/m. An abdominal (manual) thrust is applied in conjunction with the negative pressure (exsufflation) to further increase cough.
  Interventions: Behavioral: Manual and mechanical assisted cough
- Incentive spirometry (Active Comparator): The active control group will consist of individuals assigned to the oximetry with incentive spirometry group. These individuals will be given a pulse oximeter and an incentive spirometer (AirLife Company) and taught how to use them.
  Interventions: Behavioral: Incentive spirometry

INTERVENTIONS:
Behavioral: Manual and mechanical assisted cough — Individuals will be given a pulse oximeter and taught both manually assisted and mechanically assisted coughing techniques to maximize their cough. Manually assisted coughing consists of air stacking to deep insufflations. An abdominal thrust is then applied upon glottic opening to augment the cough. These subjects will also have rapid access to a mechanical in-exsufflator (CoughAssistTM) and will be trained on how to access and use this device. Mechanically assisted coughing (MAC) involves the use of the CoughAssistTM to expand the lungs and then quickly reverse the pressure to rapidly empty the lungs with expiratory (cough) flows of 600 L/m. An abdominal (manual) thrust is applied in conjunction with the negative pressure (exsufflation) to further increase cough.
  Other Names: CoughAssistTM; In-exsufflator
  Arms: Manual and mechanical assisted cough
Behavioral: Incentive spirometry — These individuals will be given a pulse oximeter and an incentive spirometer (AirLife Company) and taught how to use them.
  Other Names: spirometer
  Arms: Incentive spirometry

SUMMARY:
It is known that individuals with spinal cord injury are at increased risk for respiratory tract infections like pneumonia. Part of this risk is due to weakened chest and abdominal muscles that are vital to deep breathing and the ability to cough. The purpose of this study is to look at the effectiveness of two different treatments in preventing pneumonia and other respiratory problems in persons with SCI.

This is a randomized controlled trial investigating the effectiveness of two different treatments. Participants will be randomly assigned to one of the two treatment groups. They will not be told the details of the other intervention since this could influence or change their activities during the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic spinal cord injury that occurred more than 6 months ago
* An impaired ability to cough (cough peak flow less than 300 L/min)
* Oxygen saturation greater than or equal to 95% when awake and not receiving supplemental oxygen
* End-tidal carbon dioxide level less than 43 mm Hg
* Without a fever or other signs of an acute illness for the previous 2 weeks
* Able to learn the treatment protocol and have someone available at home to assist if needed to help set-up and use the equipment

Exclusion Criteria:

* Under 18 years of age
* Currently have a tracheotomy tube
* Have a history of an acute illness in the last 2 weeks
* Have lung disease as seen on chest x-ray that results in a baseline oxygen saturation decreasing below 95% during daytime hours and cannot be normalized by usual way of coughing
* Already utilizing an oximetry protocol
* Have a significant medical complication and psychiatric condition that would interfere with the conduct of the study or interpretation of the study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reductions in episodes of community acquired pneumonia (CAP) and related severe respiratory complications | 3 years

SECONDARY OUTCOMES:
Reductions in hospitalizations due to a primary diagnosis of a respiratory complications | 3 years
Duration of illness and hospitalization | 3 years
Impact of respiratory complications on quality of life and participation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Bach, M.D., Principal Investigator — University of Medicine and Dentistry - The New Jersey Medical School, Newark, N.J.; Steven Kirshblum, M.D., Principal Investigator — Kessler Institute for Rehabilitation, West Orange, N.J.; Trevor A. Dyson-Hudson, M.D., Study Director — Kessler Foundation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States